CLINICAL TRIAL: NCT03042338
Title: Evaluating the Feasibility of Central Executive Training for Children With ADHD
Brief Title: Central Executive Training for ADHD
Acronym: CET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J. Kofler, Associate Professor, Florida State University
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: R34MH102499 (NIH); R34MH102499 (NIH)
Record Dates: First submitted 2016-12-16; First posted 2017-02-03 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2018-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Central Executive Training1 (Experimental): Training tasks targeting working memory
  Interventions: Behavioral: CET: Central Executive Training
- Central Executive Training2 (Active Comparator): Training tasks targeting inhibitory control and response speed
  Interventions: Behavioral: CET: Comparison Executive Training

INTERVENTIONS:
Behavioral: CET: Central Executive Training — CET: Central Executive Training
  Arms: Central Executive Training1
Behavioral: CET: Comparison Executive Training — CET: Comparison Executive Training
  Arms: Central Executive Training2

SUMMARY:
Feasibility study of Central Executive Training (CET) for ADHD. The goal of the current project is to develop and assess the feasibility, acceptability, engagement, and usability of a novel, central executive (CE) working memory training intervention.

DETAILED DESCRIPTION:
The goal of the core study is to develop a central executive training (CET) intervention for children with attention-deficit/hyperactivity disorder (ADHD) and examine its feasibility, acceptability, engagement, and usability. This will involve early developmental work on software and treatment manuals followed by evaluation of the feasibility of enrolling, retaining, and treating ADHD children with CET. An evidence-informed intervention targeting central executive functioning in children with ADHD has the potential to result in clinically significant improvements in ADHD symptoms relative to extant behavioral treatments and capacity-based (short-term memory) training interventions. The long-term goal is to develop an efficacious and acceptable CET intervention with the potential for generalized improvements in, or normalization of, ADHD-related impairments in peer, family, and academic functioning.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-12 with principal ADHD diagnoses (via K-SADS)
* parent Behavior Assessment System for Children (BASC) Attention Problems or Hyperactivity subscale or ADHD-5 in clinical/borderline range based on age and gender
* teacher BASC Attention Problems or Hyperactivity subscale or ADHD-5 scale in clinical/borderline range based on age and gender.

Exclusion Criteria:

* gross neurological, sensory, or motor impairment, history of a seizure disorder, or psychosis, bipolar disorders, substance use, or intellectual disability disorders
* non-English speaking child or parent

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Rapport visuospatial/phonological working memory test | Approximately 10 minute task administered during a 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
  Outcome: stimuli correct

SECONDARY OUTCOMES:
Parent-reported ADHD symptoms (ADHD-5 rating scale) | Parent questionnaire requiring approximately 15 minutes to complete, administered to parent while child is completing the 3 hour post-treatment testing session occurring within 2 weeks of last intervention session

OTHER OUTCOMES:
Kaufman Test of Educational Achievement-3 (KTEA3) Reading Comprehension | Approximately 15 minute task administered during a 3 hour follow-up testing session occurring 2-4 months after last intervention session (variable time frame to account for school breaks)
  Growth scale value (GSV)
NIH List Sorting | Approximately 15 minute task administered during a 3 hour follow-up testing session occurring 2-4 months after last intervention session (variable time frame to account for school breaks)
  Assessing feasibility of this test as possible primary outcomes for follow-up trial
Teacher ADHD symptom ratings (ADHD-5 rating scale) | Teacher questionnaire requiring approximately 15 minutes to complete, mailed to teacher within 2 weeks of child's last intervention session
Inhibition test | Approximately 10 minute task administered during a 3 hour post-treatment testing session occurring within 2 weeks of last intervention session
  Stop-signal and go/no-go scores will be combined via weighted average (factor score). Divergent validity (expected to improve more in comparison condition than experimental condition).
Kaufman Test of Educational Achievement-3 (KTEA3) Listening Comprehension | Approximately 15 minute task administered during a 3 hour follow-up testing session occurring 2-4 months after last intervention session (variable time frame to account for school breaks)
  Growth scale value (GSV)
Kaufman Test of Educational Achievement-3 (KTEA3) Math Concepts and Applications | Approximately 15 minute task administered during a 3 hour follow-up testing session occurring 2-4 months after last intervention session (variable time frame to account for school breaks)
  Growth scale value (GSV)
Kaufman Test of Educational Achievement-3 (KTEA3) Reading Fluency | Approximately 15 minute task administered during a 3 hour follow-up testing session occurring 2-4 months after last intervention session (variable time frame to account for school breaks)
  Growth scale value (GSV)
Kaufman Test of Educational Achievement-3 (KTEA3) Math Fluency | Approximately 15 minute task administered during a 3 hour follow-up testing session occurring 2-4 months after last intervention session (variable time frame to account for school breaks)
  Growth scale value (GSV)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03042338/Prot_SAP_000.pdf